CLINICAL TRIAL: NCT03629769
Title: Effects of Proxelan Somministration in Patients With Chronic Prostatitis Cat. IIa NIH: Pilot Study
Brief Title: Effects of Proxelan Somministration in Patients With Chronic Prostatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Riccardo Bartoletti, Professor, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1103 / 2016
Record Dates: First submitted 2018-05-23; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Chronic Prostatitis; Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Premature Ejaculation
Keywords: Prostate inflammation; CPS/CPPS; Prostatitis; Proxelan
MeSH Terms: conditions — Prostatitis; Premature Ejaculation | interventions — Proxelan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with prostatitis-like symptoms (Experimental): Cohort of patients with CP/CPPS (abacterial prostatitis)
  Interventions: Drug: Proxelan

INTERVENTIONS:
Drug: Proxelan — Administration of one suppository of proxelan once a day for 30 days

SUMMARY:
The purpose of the study is to determinate the antinflammatory effects of the Proxelan on a cohort of patients affected by prostatitis'like symptoms and clinical evidence of abacterical prostatistis, trough a significative improvements of pain symptoms according to the NIH-CPSI questionnaire items, spermatozoa motility/concentration variations and the semen cytokines level decrease.

ELIGIBILITY:
Inclusion Criteria:

- prostatitis like symptoms for at least three months

Exclusion Criteria:

* significant post-voidal residual volume
* Meares and Stamey test suggestive for bacterial infection
* neoplasms,
* urinary stones,
* antibiotic therapy in the previous three months,
* irritable bowel syndrome,
* previous radiotherapic or chemiotherapic treatment,
* urethral stenosis,
* neurogenic bladder
* previous prostatic surgery

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health - Chronic Prostatitis Symptom (NIH-CPS) questionnaires score | 30 days
  Evaluation of pain symptoms trough NIH-CPS questionnaires' pain items (0-6). Values from 0 to 3 normal/slight symptoms; Values from 3 to 6 moderate symptoms; Values over 6 severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUP Ospedale cisanello, Pisa, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galeone G, Spadavecchia R, Balducci MT, Pagliarulo V. [The role of Proxelan in the treatment of chronic prostatitis. Results of a randomized trial]. Minerva Urol Nefrol. 2012 Jun;64(2):135-41. Italian. PMID 22617307